CLINICAL TRIAL: NCT04625075
Title: Manganese-Enhanced Magnetic Resonance Imaging of MyOcardial injuRY in COVID 19 (MEMORY- COVID)
Brief Title: Manganese-Enhanced Magnetic Resonance Imaging of MyOcardial injuRY in COVID 19 (COVID-19)
Acronym: MEMORY-COVID
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 20/NW/0249
Record Dates: First submitted 2020-11-09; First posted 2020-11-12 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Electrocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteer: Age and sex matched healthy volunteer
  Interventions: Diagnostic Test: Cardiac MRI; Diagnostic Test: Electrocardiogram (ECG); Diagnostic Test: Blood samples
- COVID-19 with myocardial injury: Patients hospitalised with severe COVID-19 infection and evidence of myocardial. Involvement: elevation of plasma cardiac troponin concentration (>99th centile of the upper reference limit), abnormalities on electrocardiography or abnormal echocardiography. Some patients will have suspected myocarditis or takotsubo cardiomyopathy. We will identify subgroups of interest who have left/right ventricular systolic dysfunction ± regional wall motion abnormalities, on echocardiography.
  Interventions: Diagnostic Test: Cardiac MRI; Diagnostic Test: Cardiac CT; Diagnostic Test: Electrocardiogram (ECG); Diagnostic Test: Blood samples
- COVID-19 without myocardial injury: Patients hospitalised with severe COVID-19 infection but without known elevation of plasma cardiac troponin concentration, clinically significant ECG abnormalities or an abnormal echocardiogram.
  Interventions: Diagnostic Test: Cardiac MRI; Diagnostic Test: Cardiac CT; Diagnostic Test: Electrocardiogram (ECG); Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Cardiac MRI with gadolinium and manganese contrast
Diagnostic Test: Cardiac CT — Cardiac CT to assess coronaries
  Groups: COVID-19 with myocardial injury; COVID-19 without myocardial injury
Diagnostic Test: Electrocardiogram (ECG) — ECG to assess rhythm
Diagnostic Test: Blood samples — renal function liver function full blood count, hematocrit glucose

SUMMARY:
Our understanding of the clinical manifestations of COVID-19 is growing on a daily basis and there is evidence that increased age, cardiovascular risk factors and cardiac comorbidity are strongly associated with poor outcomes. Furthermore, myocardial injury occurs and is associated with a much worse outcome and rapid increase in mortality. There have been several reports of myocarditis and heart failure following infection. The mechanisms of myocardial injury and its consequences are not well understood.

In an ongoing peer-reviewed and funded study, the investigators are evaluating the use of magnetic resonance imaging (MRI) to characterise and to understand the mechanisms of heart failure and myocarditis. Following strong encouragement by the British Heart Foundation, the investigators now propose to extend this investigation to patients who have recovered from COVID-19 infection to understand the mechanisms of myocardial injury that they have experienced. Using gadolinium and manganese-enhanced MRI combined with Computed tomography coronary angiography (CTCA), the investigators will assess the mechanisms and direct impact of myocardial injury in patients who have recovered from COVID-19 infection. This will help the investigators understand how best to manage individuals who demonstrate evidence of myocardial injury and potentially provide insights that could lead to novel treatment interventions to reduce such injury and improve patient outcomes.

DETAILED DESCRIPTION:
COVID-19 Pandemic This is the first major pandemic the modern world has faced since the Spanish Flu in 1918, with a profound impact on all aspects of society as we know it. Governments worldwide have put in place emergency plans to help tackle and reduce the rapid spread of the infection, with social isolation being implemented by most to varying degrees. As expected, healthcare systems are facing unprecedented challenges and real-time re-structuring. As well as focusing on the identification and management of critically unwell COVID-19 patients, healthcare organisations have the responsibility of protecting the public from infection and to continue the treatment of non COVID-19 related conditions. This has resulted in a complete reorganisation in how we deliver care, prioritising safety and infection control measures. In reality, this means cancelling routine clinics and procedures and has the potential to have a great impact on patient care.

COVID-19 The pool of evidence regarding this novel strain of coronavirus and the associated infection is growing as the condition unfolds. The current estimated case fatality rate varies between 1.4%-2.3%, with higher rates in the elderly, certain ethnic groups and those with co-morbidities. The largest case series from the Chinese Centre of Disease Control and Prevention reported 72,314 case records from suspected and confirmed cases. The clinical severity was reported as mild in 81.4%, severe in 13.9% and critical in 4.7%. Although clinical presentation of COVID-19 can be variable, most commonly symptoms resemble those of other viral respiratory tract infections: fever, cough, dyspnoea, myalgia and fatigue. In severe cases, COVID-19 is associated with bilateral pneumonia, acute respiratory distress syndrome (ARDS), and septic and cardiogenic shock, with higher mortality and morbidity seen in elderly and comorbid patients.

Patients with known cardiovascular risk factors or established cardiac problems are at higher risk of contracting severe acute respiratory syndrome- coronavirus-2 (SARS-CoV-2), and this confers a worse prognosis in COVID- 19 infection. It is difficult to establish the true link between COVID-19 and prevalence of cardiovascular complications due to the lack of testing in community and the cohort of patients who are admitted to secondary care, who are likely to be older and have co-morbidities and therefore are more likely to have pre-existing cardiac conditions and develop new cardiovascular complications.

COVID-19: Myocardial Injury Myocardial injury with necrosis can occur with and without overt ischaemia from acute myocardial infarction and is defined as an elevated plasma cardiac troponin concentration above the 99th centile. There are different mechanisms underlying acute myocardial injury; with ischaemia from an acute coronary syndrome and prolonged myocardial oxygen demand/supply imbalance being the most familiar. It is well recognised that an acute myocardial injury may occur in the absence of ischaemia due to a variety of cardiac and non-cardiac causes. Furthermore, this can be seen in critically unwell patients of varying aetiology and is a marker of poor prognosis.

Therefore determining the underlying mechanism is vital in guiding clinical care and improving outcomes. Myocardial injury is increasingly recognised in COVID-19 patients and, as anticipated, it correlates with severe cases and poor outcomes.5 In a cohort of 191 patients with confirmed COVID-19, plasma cardiac troponin concentrations were elevated in non survivors compared to survivors: 46% (23/50) compared to 1% (1/95) mortality.

Studies have demonstrated that rates of in-hospital death were 80 times higher in patients with myocardial injury. Interestingly temporal change in cardiac troponin showed a marked increase over time in those who did not survive, with no change on serial testing in survivors, suggestive of a progressive process of evolving myocardial injury. The mechanism of myocardial injury is not understood and it is likely that it has a similar non-direct mechanism of injury similar to that of other severe respiratory illnesses. Other putative mechanisms include direct myocardial injury due to endothelial dysfunction or cytokine release, stress cardiomyopathy, or the results of a profound ongoing myocardial oxygen supply or demand imbalance.

COVID-19: Myocardial Infarction Based on current disease patterns, COVID-19 will have a significant impact directly and indirectly on cardiovascular health. Though myocardial injury can affect those with and without cardiovascular risk factors, patients with underlying cardiac conditions are predisposed to COVID-19 and have poorer prognosis. No published cases of acute coronary syndromes have yet been described in the COVID-19 population. However, previous studies have shown that the risk of an acute myocardial infarction was higher in those with influenza and non-influenza (coronavirus) viruses. The management of acute coronary syndrome is likely to be streamlined in the face of competing clinical demands. and act upon these findings.

COVID-19: Myocarditis, stress cardiomyopathy and heart failure Previous studies demonstrated cases of acute myocarditis in Middle East Respiratory Syndrome with the use of cardiac magnetic resonance imaging. A small number of case reports have suggested fulminant myocarditis may occur in patients with COVID-19 in the setting of high viral load with autopsy findings of inflammatory mononuclear infiltrate in myocardial tissue. Among 68 deaths in a case series of 150 patients with COVID- 19, 7% were attributed to myocarditis with circulatory failure and in 33% of cases myocarditis may have played a contributing role to the patient's demise. There have been reports of COVID-19 mimicking an ST elevation myocardial infarction (STEMI), with normal coronaries and left ventricular systolic dysfunction suggesting a pattern of insult similar to that of stress cardiomyopathy. Zhou and colleagues reported that heart failure was observed in 23.0% of patients with COVID-19 presentations. Notably, heart failure was more commonly observed than acute kidney injury in this cohort and was more common in patients who did not survive the hospitalisation compared to those who did survive (51.9% vs. 11.7%). Whether heart failure is most commonly due to exacerbation of pre-existing left ventricular dysfunction versus new cardiomyopathy (either due to myocarditis or stress cardiomyopathy) remains unclear.

As this situation evolves, so will our strategies for assessment and treatment, with the use of focused bedside echocardiography and the consideration of systemic thrombolysis therapy. It is certainly possible that this will have an impact on clinical outcomes. There will be many lessons learned from this global emergency, lessons which have the potential to improve the efficiency of healthcare delivery in the future.

However, there is also a risk of worsening outcomes in conditions where there is a strong evidence base for treatment improving outcomes.

Magnetic Resonance Imaging with Late gadolinium enahancement Cardiac imaging using magnetic resonance imaging with late gadolinium enhancement is the gold-standard method for non-invasive characterisation of myocardial function and scar formation. It has been used to determine the presence of scar formation following myocardial infarction and cardiomyopathies, and has been an invaluable tool for precisely defining cardiac performance and disease.

Manganese - enhanced magnetic resonance imagining Manganese, one of the first magnetic resonance imaging contrast agents, is a calcium analogue that is taken up actively by voltage-gated calcium channels in viable myocardium. This unique property allows direct quantification of viable cardiomyocytes. The investigators have recently demonstrated that the manganese-based contrast medium, mangafodipir, is taken up by normal viable myocardium but is absent in infarcted non-functional myocardium in patients with acute myocardial infarction. In separate studies, the investigators have also shown that patients with dilated cardiomyopathy have reduced and impaired manganese uptake and this correlates with the severity of left ventricular dysfunction. Thus manganese-enhanced magnetic resonance imaging is a unique method of assessing myocardial calcium handling to detect overt or subclinical evidence of myocardial dysfunction.

Computed tomography coronary angiography. CTCA has excellent sensitivity for detecting coronary artery disease and plaque burden, both of which are associated with adverse coronary events. Furthermore, with the vast choice of cardiac imaging available, major guidelines advocate the use of CT coronary angiography as the investigation of choice for the assessment of the presence of coronary artery disease.

Rationale for Study The investigators wish to explore the cardiac consequences of severe COVID-19 infection using cardiac magnetic resonance imaging (both gadolinium and manganese enhancement) to characterise the early injury and subsequent recovery of the heart.

Furthermore, the investigators will use CT coronary angiography to determine the extent of concomitant coronary artery disease since this is likely to be the single biggest modifier of the extent of myocardial injury consequent on severe COVID-19 infection.

Study Aims There is growing evidence that myocardial injury is seen in a large number of patients with COVID-19 infections. Although there have been cases of patients infected by COVID-19 presenting with heart failure, it remains unknown whether this is a result of myocarditis, stress cardiomyopathy, acute coronary syndrome, coronary heart disease or myocardial injury related to multi-organ failure. As a result, the underlying mechanism, immediate treatment and long-term impact remains unknown. This study will improve our understanding of the underlying mechanisms which lead to myocardial injury seen in patients infected with COVID-19. This will change the way patients are treated both during the acute COVID-19 infection and in the longer term.

ELIGIBILITY:
Inclusion Criteria:

* All subjects to be entered must:

  * ≥ 18 years of age
  * if female, be non-pregnant as evidenced by a urine pregnancy test or postmenopausal or surgically sterile
  * provide written informed consent after having received oral and written information about the study

Exclusion Criteria:

have a positive pregnancy test

* women who are breast feeding
* have a history of ongoing drug abuse or alcoholism
* have a history of torsades or prolonged QT/QT corrected interval
* high degree atrioventricular block (AVB, second or third degree)
* atrial fibrillation or flutter
* have New York Heart Failure Association (NYHA) Grade IV heart failure
* have abnormal liver function tests (> x3 ULN) or a history of liver disease
* have a baseline estimated glomerular filtration rate (eGFR) (of <30 mL/min/1.73 m2)
* have uncontrolled hypertension (systolic blood pressure >200 mmHg)
* have any contraindications to MRI, including implanted devices/pacemakers
* be maintained on either a calcium channel blocker or digoxin
* known diagnosis of pheochromocytoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient cohort:
  Patients admitted to hospital with COVID-19 with and without myocardial injury
  Healthy volunteer:
  Age and sex matched healthy control with no evidence/symptoms of COVID-19
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
MRI with gadolinium | 2 years
  Measure late gadolinium enhancement
Extra-cellular volume (ECV) | 2 years
  Measure T1 values to calculate ECV (%)
Manganese MRI | 2 years
  Measure manganese uptake
CTCA | 2 years
  Measure degree of coronary disease

SECONDARY OUTCOMES:
Cardiac biomarkers | 2 years
  measure troponin profile in patients
Electrocardiogram | 2 years
  ECG Rhythm
Electrocardiogram | 2 years
  ECG ST segment
Electrocardiogram | 2 years
  ECG Rate
Electrocardiogram | 2 years
  ECG T wave morphology
Electrocardiogram | 2 years
  ECG QT interval

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be directly shared with other researchers. Anonymised MRI data will be shared with Leeds university for a central MRI database of all COVID-19 patients.

REFERENCES:
- [Derived] Singh T, Kite TA, Joshi SS, Spath NB, Kershaw L, Baker A, Jordan H, Gulsin GS, Williams MC, van Beek EJR, Arnold JR, Semple SIK, Moss AJ, Newby DE, Dweck M, McCann GP. MRI and CT coronary angiography in survivors of COVID-19. Heart. 2022 Jan;108(1):46-53. doi: 10.1136/heartjnl-2021-319926. Epub 2021 Oct 6. PMID 34615668